CLINICAL TRIAL: NCT03436485
Title: Safety and Pharmacokinetics of ODM-208 in Patients With Metastatic Castration-resistant Prostate Cancer
Acronym: CYPIDES
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3124001
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer Metastatic
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- ODM-208 Part 1 Dose escalation (Experimental)
  Interventions: Drug: ODM-208
- ODM-208 Part 2 Dose expansion (Experimental)
  Interventions: Drug: ODM-208
- ODM-208 Part 2 Drug drug interaction (Experimental)
  Interventions: Drug: ODM-208; Drug: Midazolam

INTERVENTIONS:
Drug: ODM-208 — co-administered with glucocorticoid and fludrocortisone, orally daily
Drug: Midazolam — orally
  Arms: ODM-208 Part 2 Drug drug interaction

SUMMARY:
The purpose of this first-in-man study is to evaluate safety and tolerability of ODM-208 in patients with metastatic castration-resistant prostate cancer.

DETAILED DESCRIPTION:
Safety and tolerability profile of ODM-208 will be explored

ELIGIBILITY:
Main Inclusion Criteria:

* Written informed consent (IC) obtained.
* Male aged ≥ 18 years.
* Histologically confirmed adenocarcinoma of the prostate.
* Castration resistant prostate cancer with serum testosterone < 50 ng/dl.
* Metastatic disease.
* Ongoing androgen deprivation therapy with GnRH analogue or antagonist, or have had bilateral orchiectomy.
* Received at least one prior line of novel hormonal androgen receptor (AR) targeted therapy (e.g. abiraterone, enzalutamide).
* ECOG performance status 0-1.
* Adequate marrow, liver and kidney function.
* Able to swallow study treatment.
* Part 1: Treatment with at least 1 line of chemotherapy or ineligibility for chemotherapy. Part 2: Treatment with at least 1 line of taxane-based chemotherapy in castration-sensitive prostate cancer (CSPC) or in CRPC.

Main Exclusion Criteria:

* History of pituitary or adrenal dysfunction.
* Known brain metastases or active leptomeningeal disease.
* Active infection or other medical condition that would make corticosteroid contraindicated.
* Poorly controlled diabetes.
* Hypotension or uncontrolled hypertension.
* Clinically significantly abnormal serum potassium or sodium level.
* Active or unstable cardio/cerebro-vascular disease including thromboembolic events.
* Prolonged QTcF interval.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Within first 28 days of treatment
  Highest dose level at which under 33% of patients in a cohort experience DLT

CONTACTS AND LOCATIONS:
Overall Officials: Karim Fizazi, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (20):
- United States (4):
  - University of Maryland Marlene and Stewart Greenebaum Cancer Center, Baltimore, Maryland
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - University at Buffalo, Kaleida Health Great Lakes Cancer Care Collaborative, Buffalo, New York
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Hospital, Tampere
- France (6):
  - Institute Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - Institute Paoli-Calmettes, Marseille
  - Institut de cancérologie Strasbourg Europe, Strasbourg
  - Hopital Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- United Kingdom (8):
  - The Rutherford Cancer Centre, North East, Bedlington
  - Velindre Cancer Centre, Cardiff
  - The Beatson West of Scotland Cancer Centre, Glasgow
  - The Rutherford Cancer Centre, North West, Liverpool
  - Royal Marsden Hospital, London
  - Charing Cross Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Preston Hospital, Preston

REFERENCES:
- [Derived] Fizazi K, Bernard-Tessier A, Roubaud G, Utriainen T, Barthelemy P, Flechon A, van der Voet J, Gravis G, Ratta R, Jones R, Parikh O, Tanner M, Antonarakis ES, Baldini C, Peters N, Garratt C, Ikonen T, Pohjanjousi P, Joensuu H, Cook N. Targeted Inhibition of CYP11A1 in Castration-Resistant Prostate Cancer. NEJM Evid. 2024 Jan;3(1):EVIDoa2300171. doi: 10.1056/EVIDoa2300171. Epub 2023 Dec 26. PMID 38320513